CLINICAL TRIAL: NCT06714500
Title: Transcatheter Tricuspid Valve Replacement Using the Lux-Valve Plus System for Patients With No Other Interventional Option: A Compassionate Use Study
Brief Title: Transcatheter Tricuspid Valve Replacement Using the Lux-Valve Plus System
Acronym: LuxValve
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Principle Investigator, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.029
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: LuxValve PLlus

INTERVENTIONS:
Device: LuxValve PLlus — The LuX-Valve (Jenscare Biotechnology) is a radial force-independent orthotopic TTVR device. The feasibility and efficacy of this device have been reported by several studies (11-13). However, this valve was implanted through right atrial access, where a small incision of the right chest and right atrium is needed. The LuX-Valve Plus valve replacement system is the second-generation version of the LuX-Valve and can be implanted through the jugular vein.

SUMMARY:
Tricuspid regurgitation (TR) is a common disease, and the tricuspid valve (TV) is no longer a "forgotten valve". Open heart surgery for isolated TR is uncommonly performed due to high operative risk (8-10% mortality). However, TR is associated with increased morbidity and mortality. There exists an unmet clinical need for less invasive intervention to treat TR. Transcatheter edge to edge repair (TEER) is a technique that is shown to be safe and effective in TR reduction and is associated with significant symptom improvement. However, a significant portion of TV anatomy are not suitable to be treated with TEER (e.g. coaptation gap >10mm). A wide variety of technologies has been developed in recent years. Transcatheter tricuspid valve replacement (TTVR) is one of the more promising option for tricuspid regurgitation (TR) patients at high risk for surgery. A previous study reported that transcatheter tricuspid devices, which were employed with the radial force between the device and tricuspid annulus, were radial force-dependent. However, this radial force for valve fixation may cause complications, such as conduction block and right coronary artery impingement. The LuX-Valve (Jenscare Biotechnology) is a radial force-independent orthotopic TTVR device. The feasibility and efficacy of this device have been reported by several studies. However, this valve was implanted through right atrial access, where a small incision of the right chest and right atrium is needed. The LuX-Valve Plus valve replacement system is the second-generation version of the LuX-Valve and can be implanted through the jugular vein. The first-in-human implantation was recently performed. The study aims to assess the feasibility, safety and efficacy outcome of the Lux Valve Plus system in a cohort of otherwise no surgical option patients with severe symptomatic tricuspid regurgitation despite optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50- to 90-year-old
* Severe symptomatic tricuspid regurgitation (NYHA III-IV) despite optimal medical therapy
* Deem high risk for tricuspid valve surgery determined by a multidisciplinary heart team (including cardiologists, cardiac surgeons and cardiac anesthetists)
* Anatomically not feasible with other transcatheter tricuspid valve therapy that is commercially available in Hong Kong (i.e. TriClip System)
* Capacity to provide informed consent

Exclusion Criteria:

* Systolic pulmonary artery pressure (sPAP) > 60 mmHg assessed by echocardiography
* Left Ventricular Ejection Fraction (LVEF) <40%
* Evidence of intracardiac mass, thrombus or vegetation
* Anatomical structures precluding proper device deployment or device vascular access, evaluated by echo or CT
* Surgical correction is indicated for other concomitant valvular disease (e.g., severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation); Subjects with concomitant valvular disease may treat their respective valve first and wait 2 months before being reassessed for the trial.
* Sepsis or active endocarditis within 3 months, or infections requiring antibiotic therapy within 2 weeks prior to the planned procedure
* Active peptic ulcer or active gastrointestinal (GI) bleeding precluding anticoagulation or antiplatelet therapy
* Subjects currently participating in another clinical trial of an investigational drug or device that has not yet completed its primary endpoint.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint of Major Adverse Event (MAE) | 1 year post-op
  A composite endpoint of Major Adverse Event (MAE) at 30 days post procedure: Cardiovascular Mortality, Myocardial Infarction (MI), Stroke, New onset renal failure requiring unplanned dialysis or renal replacement therapy, Severe Bleeding (includes fatal, life-threatening and extensive bleeding as defined by VARC), Non-selective tricuspid valve surgery or transcatheter re-intervention post procedure, Major cardiac structural complications, Major access site and vascular complications, New pacemaker implantation due to AV block

SECONDARY OUTCOMES:
Acute Device Success Rate | At the end of Procedure
  successful deployment of the device and removal of the delivery system as planned, with no unplanned surgery related to the device or access procedure.
Procedural Success Rate | At the end of Procedure
  Device success without clinically significant PVL, as determined by the Echo Core Lab (ECL) assessment of a discharge TTE. Subjects who die or undergo tricuspid valve surgery before discharge are procedure failures.
All-cause mortality | 30-day and 1-year post-op
  30-day and 1-year all-cause mortality
Heart failure hospitalization | 30-day and 1-year post-op
  30-day and 1-year Heart failure hospitalization
NYHA Functional Class | 30-day and 1-year post-op
  NYHA Functional Class 2. Distance of 6-Minute Walk Test (6MWT) 3. Kansas City Cardiomyopathy Questionnaire (KCCQ)：Scores are transformed to a range of 0-100, in which higher scores reflect better health status
Distance of 6-Minute Walk Test | 30-day and 1-year post-op
  Distance of 6-Minute Walk Test in meters
Kansas City Cardiomyopathy Questionnaire | 30-day and 1-year post-op
  Kansas City Cardiomyopathy Questionnaire (KCCQ)：Scores are transformed to a range of 0-100, in which higher scores reflect better health status
TR Severity | Baseline, day 1, day 30, 6-month, 1-year
  TR Severity assessed by echocardiography
Mean Tricuspid valve inflow gradient | Baseline, day 1, day 30, 6-month, 1-year
  Mean Tricuspid valve inflow gradient assessed by echocardiography
Right Atrial Volume | Baseline, day 1, day 30, 6-month, 1-year
  Right Atrial Volume assessed by echocardiography
TAPSE | Baseline, day 1, day 30, 6-month, 1-year
  TAPSE assessed by echocardiography
Right ventricular functions assessments | Baseline, day 1, day 30, 6-month, 1-year
  Right ventricular functions assessments assessed by echocardiography
Right ventricular functions assessments: fractional area change（FAC） | Baseline, day 1, day 30, 6-month, 1-year
  Right ventricular functions assessments: fractional area change（FAC）assessed by echocardiography
Right ventricular functions assessments: systolic tricuspid lateral annular tissue velocity S' | Baseline, day 1, day 30, 6-month, 1-year
  Right ventricular functions assessments: systolic tricuspid lateral annular tissue velocity S' assessed by echocardiography
Right ventricular functions assessments: Hepatic vein flow reversal | Baseline, day 1, day 30, 6-month, 1-year
  Right ventricular functions assessments: Hepatic vein flow reversal assessed by echocardiography
Systolic pulmonary artery pressure | Baseline, day 1, day 30, 6-month, 1-year
  Systolic pulmonary artery pressure assessed by echocardiography
Left Ventricular Ejection Fraction (LVEF) | Baseline, day 1, day 30, 6-month, 1-year
  Left Ventricular Ejection Fraction (LVEF) assessed by echocardiography
Paravalvular leak severity | Baseline, day 1, day 30, 6-month, 1-year
  Paravalvular leak severity assessed by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Kent So, PI, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared